CLINICAL TRIAL: NCT04168177
Title: Bilateral Erector Spinae Plane Block in Paediateric Cardiac Surgery, Randomized Study
Brief Title: Bilateral Erector Spinae Plane Block in Paediateric Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, lecturer of anaesthesia and pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ASDF
Record Dates: First submitted 2019-02-20; First posted 2019-11-19 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Intervention Model Description: patients will be randomly assigned into one of two groups, control group will receive patient controlled analgesia, and intervention group will receive ESP Block .
Who Masked: Care Provider, Outcomes Assessor
Masking Description: the data collector will be unaware of the nature of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator)
  Interventions: Procedure: PCA
- ESP Group (Active Comparator)
  Interventions: Procedure: ESP

INTERVENTIONS:
Procedure: PCA — Patient controlled analgesia
  Arms: control group
Procedure: ESP — erector spinae plane block
  Arms: ESP Group

SUMMARY:
ultrasound guided erector spinae plane block will be done for childern under going midline sternotomy for cardiac surgery. It is a novel block which is suspected to give powerful analgesia, decrease anaesthetic consumption and decrease awareness on cardiac bypass

ELIGIBILITY:
Inclusion Criteria:

* elective surgery
* childern between 4 and 10 years

Exclusion Criteria:

* emergency
* infection at injection site
* allergy to local anaestheics

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-02-17 (Actual); Primary Completion 2020-07-17 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
visual analogue score | 48 hours
  pain scores will be assessed by anaesthesia and ICU nurse. zero mean no pain an 10 indicate the worst pain.

SECONDARY OUTCOMES:
intraoperative anaesthetic consumption | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No